CLINICAL TRIAL: NCT00635635
Title: Guided Imagery for Military Sexual Trauma-Related PTSD
Brief Title: Guided Imagery for Military Sexual Trauma-Related Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Jennifer L. Strauss, PhD, Duke University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Pro00001282
Record Dates: First submitted 2008-03-09; First posted 2008-03-14 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Stress Disorder, Post Traumatic; Military Sexual Trauma
Keywords: Stress Disorders, Post-Traumatic; Anxiety,; Depression,; Guided Imagery; Military Sexual Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Military Sexual Trauma; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Guided Imagery Audio
  Interventions: Behavioral: Guided Imagery Audio
- 2 (Active Comparator): Music Audio
  Interventions: Behavioral: Music Audio

INTERVENTIONS:
Behavioral: Guided Imagery Audio — Guided Imagery Audio listened to 5x per week
  Arms: 1
Behavioral: Music Audio — Music only audio to be listened to 5x per week
  Arms: 2

SUMMARY:
Military sexual trauma (MST) is a significant women's mental health issue. There is a crucial need for effective therapies for MST-related posttraumatic stress disorder (PTSD) that are well-tolerated and can be flexibly administered in a variety of treatment settings. Guided imagery is a novel, transportable intervention technique that meets these requirements and warrants research in PTSD. The proposed study will be a randomized controlled trial of the Guided Imagery for Trauma (GIFT) intervention for women veterans with MST-related PTSD. This minimal contact intervention is designed to increase coping, affect management and relaxation skills, and to fostering more positive images and beliefs associated with surviving trauma. The feasibility and tolerability of GIFT have already been demonstrated in an open-label pilot of 15 women veterans with MST-related PTSD, with very promising initial results.

DETAILED DESCRIPTION:
Study Aims: The primary aims of this study are: (1) To determine the efficacy of the GIFT intervention for women veterans with MST-related PTSD. (2) To determine the effects of GIFT on mental health and health services utilization, and neurobiological outcomes. (3) To identify predictors of GIFT treatment outcomes.

Research Plan: We will conduct a 12-week randomized, controlled trial of GIFT in 38 women veterans with MST-related PTSD. Half will be randomly assigned to GIFT and half to a music control group. GIFT includes a pretreatment orientation and midpoint consultation session with a clinician facilitator, a guided imagery audio, daily self-monitoring of audio use, and weekly telephone coaching calls with the facilitator. The music control condition is designed to control for all nonspecific aspects of GIFT and matches the GIFT protocol in all ways but the two specific "ingredients" through which GIFT is hypothesized to have its effect: (1) the guided imagery audio, and (2) the facilitator's help in structuring and focusing use of the guided imagery audio. Thus, the key differences between the two groups are that controls will receive an audio of the relaxing background music used on the guided imagery audio, but not the guided imagery exercises, and controls' contacts with the facilitator is limited to psychoeducational information and general support, and will not include help in structuring and focusing use of the audio, which is a key component of GIFT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Status as a women veteran
3. Receives care at the Durham VAMC
4. History of MST, confirmed by CAPS interview
5. DSM-IV diagnosis of PTSD, confirmed by CAPS interview
6. Able to participate in a research interview in English.
7. Regular telephone access

Exclusion Criteria:

1. Current diagnosis of organic, psychotic, or bipolar disorder
2. Suicidality or parasuicidality
3. Ongoing family violence
4. Alcohol or drug abuse within previous 3 months
5. Enrolled in cognitive-behavioral/exposure-based therapy for PTSD during study period. Supportive therapy and some psychiatric medications (if stabilized at least 3 months prior to enrollment) are acceptable. Although patients may use medications, no new medications will be started during the study. This includes, but is not restricted to, SSRIs, benzodiazepines, barbiturates, antiepileptic drugs, antidepressants, buspirone, non-benzodiazepine hypnotics, stimulants, or antipsychotics.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
PTSD Severity - Clinician Administered PTSD Scale (CAPS) | Midpoint and Endpoint

SECONDARY OUTCOMES:
Neuroactive Steroid assay | Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Strauss, PhD, Principal Investigator — Duke University
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States